CLINICAL TRIAL: NCT02301377
Title: Exploring Novel Interventions to Improve Adherence in Children With Cystic Fibrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Aarti Shakkottai, Clinical Fellow, Division of Pediatric Pulmonology, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HUM00080071
Record Dates: First submitted 2014-11-21; First posted 2014-11-25 (Estimated); Results first posted 2015-07-16 (Estimated); Last update posted 2015-07-16 (Estimated); Status verified 2015-06

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention Group (Active Comparator): Participants will receive a Spiro PD personal spirometer that will allow them to measure their lung function at home and provide medication reminders. Participants will be instructed to use the device to check their lung function once a week. They will also be asked to use the medication reminder feature of their device daily. Participants in this group will receive a telephone call once a week from the research team to review lung function results and answer questions. All participants need to fill out a quality of life questionnaire at the time of enrollment and at the end of the study. Participants will be asked to sign a release form so their pharmacies can be contacted for prescription refill data to monitor adherence over the course of the study. All participants will be asked to come to their quarterly clinic visits with their pediatric pulmonologist where their height, weight, body mass index, lung function and frequency of hospitalizations will be assessed.
  Interventions: Device: Spiro PD personal spirometer
- Control (No Intervention): Participants will be asked to fill out a quality of life questionnaire at the time of enrollment and at the end of the study. All participants will be asked to come to their quarterly clinic visits with their pediatric pulmonologist where their height, weight, body mass index, lung function and frequency of hospitalizations will be assessed. All participants will be asked to sign a release form so their pharmacies can be contacted for prescription refill data to monitor adherence over the course of the study.

INTERVENTIONS:
Device: Spiro PD personal spirometer
  Arms: Intervention Group

SUMMARY:
The investigators know that adherence to medications in children with cystic fibrosis (CF) is poor. Forgetfulness has often been reported as a barrier to adherence by both CF patients and their parents. Many of the investigators patients also report being motivated by the results of their lung function studies (PFTs) to stay adherent to their medications. In this study, the investigators would like to see if providing medication reminders and allowing patients to measure their lung function at home will lead to better adherence. This will be a pilot study to determine the feasibility of providing such as a device to children with CF.

DETAILED DESCRIPTION:
This is a randomized controlled trial to assess the impact of home lung function monitoring and medication reminders on adherence, clinical outcomes and quality of life in children with cystic fibrosis (CF) who are between 10 and 21 years of age.

Participants will be randomly assigned to either an intervention group or a control group. Those in the intervention group will receive a personal spirometer device that provides medication reminders and allows for lung function monitoring at home. The control group will receive the current standard of care. All participants will be aware that their adherence is being monitored over the course of the study using prescription refill data. Changes in lung function, body mass index and rate of hospitalization will be used as measures of clinical outcome. Responses to age-appropriate well-validated patient questionnaires will be used to assess the impact of the investigators interventions on quality of life and perceptions of treatment burden.

Since this device has never been previously studied in this patient population, the investigators would like to do a pilot study with 5 patients (3 in the intervention group and 2 in the control group) over a 3-month period to determine feasibility. This will also help us with the investigator power calculations and ultimately deciding the number of participants that will be needed for the larger study.

ELIGIBILITY:
Inclusion Criteria:

1. Age 10-21 years
2. Confirmed diagnosis of cystic fibrosis (CF) either by a sweat chloride ≥ 60mEq/L or the presence of two disease-causing mutations
3. Patients must be clinically stable with at least 1 month from their last hospitalization or use of oral antibiotics for a pulmonary exacerbation
4. Signed informed consent from the patient and/or from the parent/legal guardian, if younger than 18 years.

Exclusion Criteria:

1. Age less than 10 years or greater than 21 years
2. Clinically unstable

Ages: 10 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Actual)
Dates: Start 2014-11; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aarti Shakkottai, MD, Principal Investigator — University of Michigan; Samya Nasr, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention Group: Subjects in this group were asked to use the Spiro PD personal spirometer to check their lung function once a week for 3 months. They were also asked to use the medication reminder feature of their device daily. Participants were trained on the appropriate use of their device at the time of enrollment. They also received weekly telephone calls from a respiratory therapist to review that week's lung function results. They filled out a quality of life questionnaire at enrollment and at 3 months. Information regarding their height, weight, lung function and frequency of hospitalizations over the previous 3 months were obtained at enrollment and 3-months from review of their medical records. Pharmacies were contacted for refill data during the 3-month study duration for inhaled hypertonic saline, dornase alfa and CF multivitamins.
- Control: Subjects in this group had their adherence to inhaled hypertonic saline, dornase alfa and CF multivitamins during the 3-month study duration monitored through the use of prescription refill histories. They filled out a quality of life questionnaire at enrollment and 3 months. Their height, weight, lung function and frequency of hospitalizations over the previous 3 months was obtained at enrollment and 3-months from review of their medical records.
Period: Overall Study
Arm/Group | Intervention Group | Control
Started | 3 | 2
Completed | 3 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Control | Total
Number analyzed (Participants) | 3 | 2 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.51 (0.64) | 11.93 (1.29) | 11.67 (0.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 0 | 1 | 1
Forced expiratory volume in 1 second (FEV1) [Mean (Standard Deviation); unit: %predicted] | 74.33 (16.65) | 93 (1.41) | 81.8 (15.61)
Body Mass Index (BMI) Percentile [Mean (Standard Deviation); unit: Percentile] | 64.33 (19.14) | 41.5 (16.26) | 55.2 (20.14)
Cystic Fibrosis Questionnaire-Revised (CFQ-R) Treatment Burden Domain Score (Child) [Mean (Standard Deviation); unit: units on a scale] — This is a well-validated measure of health-related quality of life among children with CF. It assesses functionality in several disease-specific domains including treatment burden. A total score is calculated for each domain, which varies based on the number of questions in that domain. This is then converted to a scaled score between 0-100 for better comparison between the domains. Higher scores reflect better quality of life.
  units on a scale | 74.33 (6.35) | 78 (31.11) | 75.8 (16.31)
Cystic Fibrosis Questionnaire-Revised (CFQ-R) Treatment Burden Domain (Parent) [Mean (Standard Deviation); unit: units on a scale] — This is a well-validated measure of health-related quality of life among children with CF. It assesses functionality in several disease-specific domains including treatment burden. A total score is calculated for each domain, which varies based on the number of questions in that domain. This is then converted to a scaled score between 0-100 for better comparison between the domains. Higher scores reflect better quality of life.
  units on a scale | 59.33 (17.24) | 61 (24.04) | 60 (17.14)

OUTCOME MEASURES:

1. Primary Outcome: Medication Adherence
Description: Overall adherence to inhaled hypertonic saline, dornase alfa and CF multivitamins based on prescription refill data. The actual number of prescriptions of each of the three medications filled in the 3-month period was divided by the number that should have been filled based on the prescribed amount of each medication and that value was multiplied by a 100 to generate a percentage.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: Percent Adherence
Arm/Group | Intervention Group | Control
Number analyzed (Participants) | 3 | 2
Percent Adherence | 91.6 (14.43) | 100 (0)

2. Secondary Outcome: Cystic Fibrosis Questionnaire-Revised (CFQ-R)Treatment Burden Domain Score (Child)
Description: Response of the participants to the treatment burden domain of the CFQ-R at the end of 3 months
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Group | Control
Number analyzed (Participants) | 3 | 2
units on a scale | 81.66 (16.80) | 72.5 (23.33)

3. Secondary Outcome: Cystic Fibrosis Questionnaire-Revised (CFQ-R) Treatment Burden Domain Score (Parent)
Description: Response of the parents/caregivers to the treatment burden domain of the CFQ-R at the end of 3-months
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Group | Control
Number analyzed (Participants) | 3 | 2
units on a scale | 67 (19.05) | 66.5 (31.82)

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Intervention Group | Control
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/2
Other Adverse Events (participants affected / at risk) | 0/3 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes